CLINICAL TRIAL: NCT02620345
Title: Uterine Fibroids Are a Very Common Finding in Women of Reproductive Age. Ready Safety Study Dydrogesterone + Multivitamin Nature in Women of Reproductive Age and Women Pregnancy
Brief Title: Fibroids in Women of Reproductive Age and Women Pregnancy
Acronym: Fibroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trieu, Nguyen Thi, M.D. (Individual)
Responsible Party: Principal Investigator, Triệu, Nguyễn Thị, M.D., Clinical Study, Trieu, Nguyen Thi, M.D.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dydrogesterone Multivitamin
Record Dates: First submitted 2015-11-14; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Fibroids
Keywords: Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dydrogesterone M/ Women Pregnancy (Experimental): * Reducing the size of fibroids with medication
  * Drug: Dydrogesterone M 15mg/Fibroids/Women Pregnancy
  * Dosage:
  * 1tablet/24 hours/day/ (when seeing fibroids to 4 weeks after postpartum). Dydrogesterone 15mg/day Beta Carotene 4000 IU/day Ascorbic Acid 100 mg/day Cholecalciferol 400 IU/day Dl-Alpha Tocopheryl Acetate 11IU Thiamin Mononitrate 1.5 mg/day Riboflavin 1.7 mg/day Niacinamide 18 mg/day Pyridoxine Hydrochloride 2.6 mg/day Folic Acid 400 mcg/day Cyanocobalamin 4mcg/day Calcium Carbonate 150 mg/day Ferrous Fumarate 27 mg/day Zinc Oxide 25 mg/day
    * The lost in size of fibroids throughout pregnancy after 48 weeks.
  Interventions: Drug: Dydrogesterone M ( case 1 )
- Dydrogesterone M/ Reproductive Age (Experimental): * Reducing the size of fibroids with medication
  * Drug: Dydrogesterone M 15mg/Fibroids/Reproductive Age
  * Dosage:
  * 1tablet/24 hours/day/24 weeks ( from discovered fibroids through 24 weeks). Dydrogesterone 15mg/day Beta Carotene 4000 IU/day Ascorbic Acid 100 mg/day Cholecalciferol 400 IU/day Dl-Alpha Tocopheryl Acetate 11IU Thiamin Mononitrate 1.5 mg/day Riboflavin 1.7 mg/day Niacinamide 18 mg/day Pyridoxine Hydrochloride 2.6 mg/day Folic Acid 400 mcg/day Cyanocobalamin 4mcg/day Calcium Carbonate 150 mg/day Ferrous Fumarate 27 mg/day Zinc Oxide 25 mg/day
    * The lost in size of fibroids after 24 weeks.
  Interventions: Drug: Dydrogesterone M ( case 2 )

INTERVENTIONS:
Drug: Dydrogesterone M ( case 1 ) — Dydrogesterone Multivitamin nature
  * Fibroids / Women Pregnancy ( discovered fibroids during pregnancy ) Dydrogesterone Multivitamin nature.
  * 1tablet/24 hours/day (to 4 weeks after postpartum)
  Other Names: Dydrogesterone M
  Arms: Dydrogesterone M/ Women Pregnancy
Drug: Dydrogesterone M ( case 2 ) — Dydrogesterone Multivitamin nature
  * Fibroids/ Women of Reproductive age ( discovered fibroids )
  * 1tablet/24 hours/day ( from discovered fibroids through 6 months)
  Other Names: Dydrogesterone M
  Arms: Dydrogesterone M/ Reproductive Age

SUMMARY:
Dydrogesterone Multivitamin Nature treatment of fibroids in women of reproductive age and women pregnancy to lost the size fibroids.

DETAILED DESCRIPTION:
Uterine fibroids are a very common finding in women of reproductive age. But may fibroids grow in the first trimester pregnancy.

Clinically has shown that:

Uterine fibroids are associated with an Heavy or prolonged menstrual periods. Abnormal bleeding between menstrual periods.

Uterine fibroids are associated with an increased rate of spontaneous miscarriage, preterm labor, placenta abruption, malpresentation, labor dystocia, cesarean delivery, and postpartum hemorrhage, pain is the most common complication of fibroids during pregnancy. Can usually be controlled by conservative treatment on Dydrogesterone Multivitamin nature.

ELIGIBILITY:
Inclusion Criteria:

* Procedure to treatment of fibroids in pregnancy and in women desiring future fertility.

Exclusion Criteria:

* Whether or not you are having symptoms from the fibroids
* If you might want to become pregnant in the future
* The size of the fibroids
* The location of the fibroids
* Your age and you might be

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-01; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Measure of fibroid size in millimeters | from 4 weeks to 20 weeks
  * Patients fulfilling inclusion and exclusion criteria.
  * Measure to have Fibroids size > 50mm x 60mm.
    * Will be divided into two groups
  Group (A): Women Pregnancy.
  * Measure of fibroid size in millimeters < 50mm x 60mm.
  Group (B): Women Reproductive age.
  * Measure of fibroid size in millimeters < 50mm x 60mm.

SECONDARY OUTCOMES:
Measure of fibroid size in millimeters | from 20 weeks to 48 weeks
  Group (A):Women Pregnancy.
  - Measure of fibroid size in millimeters to loss the fibroids.
  Group (B): Women Reproductive age
  - Measure of fibroid size in millimeters to loss the fibroids.

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Thi Trieu, Master, Study Director — Tran Minh Duc, Dr.

REFERENCES:
- See also: Contemporary Management of Fibroids in Pregnancy — http://www.ncbi.nlm.nih.gov
- See also: What is the treatment for uterine fibroids? — http://www.medicinenet.com